CLINICAL TRIAL: NCT02857621
Title: Evaluation of Pressure Applying Efficiency in Multi-Layer Bandaging Among Physiotherapists Who Treat Lymphedema
Brief Title: Evaluation of Pressure Applying Efficiency in Multi-Layer Bandaging
Status: Completed | Type: Observational
Sponsor: Assuta Hospital Systems (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other); University of Haifa (Other)
Responsible Party: Sponsor
Other Study IDs: 2016032
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2016-06

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Lymphedema is a condition characterized by excess accumulation of protein rich tissue fluid in interstitial spaces. It is a progressive chronic disease and without appropriate management may result in serious complications. In Israel, patients are referred to physiotherapists certified in treatment for lymphedema. According to the International Society of Lymphology (ISL) the best treatment is a holistic, multidiscipline approach. Amongst the different methods of lymphedema management, the use of compression is the only treatment that has shown to be effective in randomized controlled trials.

The ISL recommends that patients with lymphedema in the lower limb ought to bandage their leg with multi-layer bandaging on a daily basis for a period of two to four weeks. A new classification system for compression bandages was recommended; pressure of <20 mmHg was categorized as mild, 20-40 mmHg as medium, 40-60 mmHg as strong and ≥60 mmHg as very strong. In patients with leg edema, bandages with strong pressure were shown to be the most effective. However, in the presence of a venous ulcer on a lymphatic leg, pressure between 35 and 45 mmHg is the widely accepted range for sufficient and safe compression. The use of measurement instruments is currently the only realistic method for determining the actual pressure achieved beneath the bandage. However, it is neither economical nor feasib¬le nor is it realistic in terms of time.

Recent studies show that many healthcare professionals use inadequate sub-bandage pressure. No study so far has focused on therapists that are trained in lymphatic treatment. In spite of correct pressure bandaging importance, the question whether physiotherapists succeed in correctly applying it is left unanswered. The main purpose of this study is to evaluate the pressure applying efficiency in multi-layer bandaging among physiotherapists in Israel who treat lymphedema.

34 physiotherapists trained in lymphatic treatment will be recruited for this research. Each volunteer will receive a questionnaire concerning their self-perceived competence in the application of compression bandages. Afterwards, two practical trials will be held a week apart in which the subjects will be asked to apply bandages using strong and medium pressure. Using PicoPress®, pressure will be measured directly after bandaging and two hours later. Our hypothesis is that the majority of therapists will properly apply medium or strong pressure on the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* Physical Therapists trained in Lymphatic treatments

Exclusion Criteria:

* Have not treated a Lymphatic patient in the past two years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physical Therapists who have been specifically trained in Lymphatic therapy and have administered these treatments in the past two years.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-08; Primary Completion 2017-04-23 (Actual); Study Completion 2017-04-23 (Actual)

PRIMARY OUTCOMES:
Sub-bandage pressure | Two hours
  Resting pressure will be measured directly after bandaging and two hours later using a PicoPress® measurement device.

CONTACTS AND LOCATIONS:
Overall Officials: Woldman Anat, BPT, Study Director — Physical Therapist at Maccabi HMO
Locations (1):
- Maccabi Healthcare Services, Bat Yam, Israel

IPD SHARING:
Plan to Share IPD: No